CLINICAL TRIAL: NCT02654678
Title: Follow-up Safety Trial in Children With Chronic Heart Failure Therapy Receiving Orodispersible Minitablets of Enalapril
Acronym: LENA-WP10
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ethicare GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-602295-03; 2015-002397-21 (EudraCT Number)
Record Dates: First submitted 2016-01-04; First posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Heart Failure; Dilated Cardiomyopathy; Congenital Heart Disease
MeSH Terms: conditions — Heart Failure; Cardiomyopathy, Dilated; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enalapril Orodispersible Minitablets (Experimental): Individually adapted dose of enalapril consisting of 1 to maximum 4 enalapril ODMTs of 0.25 mg and/or 1 mg and/or other prescribed treatment of heart failure.
  Interventions: Drug: Enalapril Orodispersible Minitablet

INTERVENTIONS:
Drug: Enalapril Orodispersible Minitablet — Weight-dependent long-term treatment scheme with enalapril ODMTs of 0.25 and/or 1 mg strength
  Other Names: Enalapril ODMT

SUMMARY:
Paediatric long-term safety follow-up clinical trial in maximum 100 children with heart failure due to dilated cardiomyopathy or congenital heart disease, from 1 day to less than 12 years of age at recruitment into the preceding short-term pharmacokinetic (PK)/pharmacodynamic (PD) trials. Pharmacodynamic measurements and renal monitoring in all children after 1 , 4, 7 and 10 months of follow-up; in addition PK assessments as well as acceptability and palatability assessments in children still under enalapril Orodispersible Minitablet (ODMT) treatment.

DETAILED DESCRIPTION:
This clinical trial is one of three clinical trials of the European Commission (FP7)-funded "LENA" (Labeling of Enalapril from Neonates to Adolescents) project: 50 children with heart failure due to dilated cardiomyopathy (LENA-Work Package (WP)08 Trial) and 50 children with heart failure due to congenital heart disease (LENA-WP09 Trial) get treated with an optimal dose of enalapril ODMTs for up to 8 weeks after thorough, individualised titration and get invited to join this 10 months Safety Follow-up Study (LENA-WP10 Trial).

Reliable data on the long-term safety of enalapril in paediatric patients are currently not available. By conducting this long-term Safety Follow-up Trial in children who received or still receive enalapril Orodispersible Minitablets at the end of the 8-weeks PK/PD LENA-Work Package (WP)08 (children with heart failure due to dilated cardiomyopathy) and LENA-WP09 (children with heart failure due to congenital heart disease) Trials using sensitive and highly specific assay methodology, it will be possible to add to the generation of reliable PK and PD data in the whole paediatric age range from birth to 12 years. In addition, this follow-up study will allow to systematically collect follow-up information over 10 more months, so in total 12 months, in paediatric patients under long-term enalapril ODMT treatment and in paediatric patients who had received at least 3 days of ODMT treatment but then stopped for any reason.

The End-of-study Visit of the WP08 and WP09 Trials is also the First Visit of the Follow-up Study. Further Visits occur after 1 month, 4 months, 7 months and 10 months.

At each Visit blood pressure and renal monitoring as well as pharmacodynamic parameters and adverse events are assessed. In children under ongoing enalapril ODMT treatment, single PK sampling as well as acceptability and palatability assessments are made at each Visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients from the WP08 and WP09 Trials who have been treated with enalapril Orodispersible Minitablets and are still under ODMT treatment.
* Patients from the WP08 and WP09 Trials who have been treated for at least 3 days with enalapril Orodispersible Minitablets and are no longer under ODMT treatment.
* Written informed consent from parent(s)/legal representative provided written informed consent for participation in this long term follow-up study and assent from the patient according to national legislation and as far as achievable from the child.

Exclusion Criteria:

Patients who have been enrolled and treated in the WP08 or WP09 Trials have fulfilled the respective in- and exclusion criteria of those protocols. As it is the aim of this Follow-up Study to observe the safety of all patients exposed to enalapril ODMT treatment, no additional exclusion criteria are defined in this protocol. However, adapted to the health situation of the patient, the investigator will decide whether planned study activities can be performed.

Ages: 8 Weeks to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Adverse Reactions | up to month 10
  Adverse Reaction definition according to European Directive 2001/20/EC, assessed at each Visit concerning intensity and causality

SECONDARY OUTCOMES:
Blood pressure | At every Visit: (day 0, month 1, 4, 7, 10)
  Measurement pre-dose after 5 minutes at rest at every Visit up to end of treatment at Month 10
Renin | Pre-dose at each Visit: (day 0, month 1, 4, 7, 10)
  Renin to assess the Renin-angiotensin-aldosterone system (RAAS) measured at every Visit up to end of treatment at Month 10
Angiotensin 1 | Pre-dose at each Visit: (day 0, month 1, 4, 7, 10)
  Angiotensin 1to assess the Renin-angiotensin-aldosterone system (RAAS) measured at every Visit up to end of treatment at Month 10
Aldosterone | Pre-dose at each Visit: (day 0, month 1, 4, 7, 10)
  Aldosterone to assess the Renin-angiotensin-aldosterone system (RAAS) measured at every Visit up to end of treatment at Month 10
Plasma Renin Activity | Pre-dose at each Visit: (day 0, month 1, 4, 7, 10)
  Plasma renin activity to assess the Renin-angiotensin-aldosterone system (RAAS) measured at every Visit up to end of treatment at Month 10
Creatinine | Pre-dose at each Visit: (day 0, month 1, 4, 7, 10)
  Creatinine for renal monitoring measured at every Visit up to end of treatment at Month 10
Urea nitrogen | Pre-dose at each Visit: (day 0, month 1, 4, 7, 10)
  Urea nitrogen for renal monitoring measured at every Visit up to end of treatment at Month 10
Serum potassium | Pre-dose at each Visit: (day 0, month 1, 4, 7, 10)
  Serum potassium for renal monitoring measured at every Visit up to end of treatment at Month 10
Brain-Natriuretic-Peptides (BNP) | Pre-dose at each Visit: (day 0, month 1, 4, 7, 10)
  BNP measured at every visit up to end of treatment at Month 10 to observe disease severity
Micro-albuminuria | Pre-dose at each Visit: (day 0, month 1, 4, 7, 10)
  Measurement of micro-albuminuria for renal monitoring measured at every Visit up to end of treatment at Month 10
Clinical haematology | Day 0 and Month 10
  Assessment at First and Last Study Visit at the end of treatment at Month 10
ECG | Day 0 and Month 10
  Assessment at First and Last Study Visit at the end of treatment at Month 10
Plasma concentration of enalapril and its active metabolite enalaprilat under long-term treatment | Pre-dose at each Visit: (day 0, month 1, 4, 7, 10)
  At each Visit in children under enalapril ODMT treatment a single blood sample will be collected to measure the enalapril and enalaprilat plasma levels during long-term treatment; population-kinetic investigation
Acceptability assessment of enalapril ODMTs | At each Visit: (day 0, month 1, 4, 7, 10)
  Acceptability assessment at each Visit up to end of treatment at 10 months in children under enalapril ODMT treatment according to an age-appropriate scale
Palatability assessment of enalapril ODMTs | At each Visit: (day 0, month 1, 4, 7, 10)
  Palatability assessment at each Visit up to end of treatment at Month 10 in children under enalapril ODMT treatment according to an age-appropriate scale

CONTACTS AND LOCATIONS:
Overall Officials: Saskia N. de Wildt, MD,PhD, Study Chair — Sophia Children's Hospital, Erasmus MC; Michiel Dalinghaus, MD,PhD, Principal Investigator — Sophia Children's Hospital, Erasmus MC; J.M.P. J. Breur, MD,PhD, Principal Investigator — Wilhelmina Children's Hospital, University Medical Center Utrecht; Ida Jovanovic, Prof,MD,PhD, Principal Investigator — Univerzitetska Dečja Klinika Belgrade; Christoph Male, Prof,MD,PhD, Principal Investigator — Medical University of Vienna; Michael Burch, Prof,MD,PhD, Principal Investigator — Great Ormond Street Hospital for Children NHS Trust London; András Szatmári, Prof,MD,PhD, Principal Investigator — Hungarian Paediatric Heart Centre, Göttsegen Gyorgy Hungarian Institute of Cardiology
Locations (6):
- Medical University of Vienna, Vienna, Austria
- Hungarian Paediatric Heart Centre,Göttsegen Gyorgy Hungarian Institute of Cardiology, Budapest, Hungary
- Netherlands (2):
  - Sophia Children's Hospital Erasmus MC, Rotterdam
  - Wilhelmina Children's Hospital, University Medical Center Utrecht, Utrecht
- Univerzitetska Dečja Klinika, Belgrade, Serbia
- Great Ormond Street Hospital for Children NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Serious Adverse Event information